CLINICAL TRIAL: NCT03900871
Title: Prospective, Randomized, Blind, Parallel Controlled Clinical Research Programme on the Effect of Aspirin on the Disease Free Survival Rate of Esophageal Carcinoma
Brief Title: Clinical Research on the Effect of Aspirin on the Disease Free Survival Rate of Esophageal Carcinoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018051702
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Aspirin as an Adjuvant Therapy, to Observe Its Effect on the Disease Free Survival Rate of Patients With Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Acetylsalicylic acid
- Control group (Placebo Comparator)
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Acetylsalicylic acid — Aspirin (aspirin), also known as acetylsalicylic acid (acetylsalicylic acid), is a salicylic acid drug commonly used as a painkiller, antipyretic and anti-inflammatory drug. There is growing evidence that aspirin has a preventive effect on certain cancers, especially gastrointestinal cancers, and that taking aspirin every day can reduce the risk of colon cancer, and in vitro experiments have also shown that aspirin inhibits the growth of a variety of cancer cells and induces apoptosis.

SUMMARY:
Esophageal cancers are the seventh most common cancer in the world and one of the most common causes of cancer deaths. In some parts of China, the incidence of SCC is among the highest in the world. Despite surgery and adjuvant radiotherapy, the prognosis for SCC patients was disappointing. There is therefore an urgent need for new prevention and treatment strategies.

Epidemiological investigations have found that about 25% of human tumors are associated with chronic inflammation caused by a variety of causes, and chronic inflammation activates nuclear transcription factors (nuclear Factor,NF), induces gene and epigenetic changes such as DNA methylation, tumor suppressor gene point mutations, and post-translational modification, and participates in the process of tumorigenesis. It has been noted that the long-term regularity of the use of non-steroidal anti-inflammatory drugs aspirin can reduce the incidence and mortality of a variety of tumors, including esophageal cancer.

Aspirin is the earliest, most extensive and common antipyretic analgesics and anti-rheumatism drugs used to play an anti-inflammatory role by inhibiting the synthesis of PGs. COX-2 is a key enzyme in the synthesis of PGs, so it is speculated that the anti-tumor effect of aspirin inhibits the PGs of COX and its inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with malignant tumors after radical operation of esophageal squamous cell carcinoma without merging other parts; Pathological results are shown as all staging; Immunohistochemical staining showed positive COX-2 expression; Aspirin or other non-steroidal anti-inflammatory drugs have not been taken in the past; No abnormalities found in coagulation function; Between the ages of 18-70 and five, gender is not limited; Patient KPS≥90, expected survival period of more than 6 months; Patient Signs Informed Consent statement; Pregnant women with fertility must be negative in pregnancy trials.

Exclusion Criteria:

* Severe coagulation dysfunction; Severe liver, kidney and cardiac dysfunction; The lesion failed to completely remove; Active digestive tract Ulcers; Reflux esophageal disease; Allergies to aspirin or other drugs containing salicylic acid; History of asthma caused by salicylic acid salts or salicylate containing substances and non-steroidal anti-inflammatory drugs; COX-2 expression of immune tissue chemical staining weak or not expressed; Wide transfer of the whole body; Ever taken aspirin or other non-steroidal anti-inflammatory drugs; Pregnant and lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-04-10 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 years
  To observe the effect of aspirin on the disease free survival of patients with esophageal squamous cell carcinoma after operations

CONTACTS AND LOCATIONS:
Overall Officials: Junfeng Liu, Study Chair — Hebei Medical University
Locations (1):
- Junfeng Liu, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No